CLINICAL TRIAL: NCT03480204
Title: Patient Status Engine (PSE): EARLY FEASIBILITY AND USABILITY STUDY
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Isansys Lifecare LTD (Unknown)
Responsible Party: Principal Investigator, Dan Cantillon, Principal Investigator, The Cleveland Clinic
Other Study IDs: 17-1656
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Arrhythmia
Keywords: Telemetry, Patch Monitor, Alarm Fatigue
MeSH Terms: conditions — Arrhythmias, Cardiac; Alert Fatigue, Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the feasibility and usability of a wearable patch as a cardiac monitor for non-ICU hospitalized patients.

DETAILED DESCRIPTION:
This study evaluates the feasibility and usability of a wearable patch cardiac monitor, gateway and server concomitant with standard-of-care cardiac telemetry monitoring for non-ICU hospitalized patients on a selected nursing ward at the Cleveland Clinic Heart and Vascular Institute. All patients will receive routine clinical care on the basis of the traditional telemetry monitoring using the usual processes. The patch monitor data will not be reviewed in real-time, and only analyzed post hoc for agreement with the standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old and able to provide informed consent
* Standard indication for cardiac telemetry monitoring (institutional standardized criteria) with valid electronic order

Exclusion Criteria:

* Cardiac implantable device (pacemaker or ICD)
* Contact precautions or isolation
* Telemetry discontinuation planned within 12 hours (i.e. anticipated discharge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-ICU hospitalized patients on the J8-3 nursing ward at the Cleveland Clinic Heart and Vascular Institute
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Connectivity | 48 hours
  Successful patch application by nursing, and transmission of cardiac waveform data to gateway and then to offline secure server
Continuity | 48 hours
  Loss of cardiac waveform signal from patch compared with traditional telemetry monitor.

SECONDARY OUTCOMES:
Agreement for cardiac arrhythmia detection (post hoc, offline) | 48 hours
  Analysis of cardiac arrhythmia detections on patch compared with traditional telemetry for agreement, concordance and discordance.
Body temperature (post hoc, offline) | 48 hours
  Body temperature recorded by patch compared with nursing documentation in a post hoc analysis. Data from patch will not be assessed for patient care in real time.
Cardiac waveform (post hoc, offline) | 48 hours
  Pre-specified analysis of cardiac waveform characteristics in association with pre-specified clinical events such as deployment of emergency response team.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cantillon, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States